CLINICAL TRIAL: NCT07088341
Title: the Role of Programmed Death Ligand 1 in Diagnosis of Colorectal Cancer
Brief Title: Role of Programmed Death Ligand 1 in Colorectal Cancer
Acronym: SPDL1
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Mamdouh Mohamed Abdellah, resident doctor, Assiut University
Other Study IDs: sPDL-1 in colorectal cancer
Record Dates: First submitted 2025-07-19; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Colo-rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — serum or plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: elisa — enzyme- linked immunesorbent assay ( ELISA ) was used to measure soluble programmed death ligand-1 level

SUMMARY:
1. - Evaluation of diagnostic importance of soluble programmed death ligand-1 in patient with recently diagnosed as Colorectal cancer at different stages of disease .
2. Correlation of SPDL-1 level and clinco-pathological data of patients at presentation .

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is a significant cause of cancer- related deaths worldwide, and its incidence and mortality are increasing each year. It accounts for approximately 10% of all annually diagnosed cancers and cancer-related deaths worldwide[1]

Most colon cancer is sporadic, and approximately 5 percent are due to an inherited genetic mutation, mostly due to Lynch syndrome (hereditary nonpolyposis colon cancer or HNPCC) and familial adenomatous polyposis (FAP). The transition from normal colon epithelium to invasive cancer takes several years and most commonly follows a sequence characterized by the accumulation of genetic mutations, adenoma formation, and subsequent carcinogenesis (adenoma-carcinoma sequence).

Programmed death-1 (PD-1) is an immunoglobulin superfamily type I transmembrane glycoprotein consisting of 288 amino acids, which is expressed on different immune cells, especially on T cells[2]. Programmed death ligand 1 (PD-L1) is one ligand of PD-1. Soluble programmed death ligand 1 (sPD-L1) is released from PD-L1-positive cells, which binds to receptor of PD-1, participates in immune regulation [2]. Furthermore, sPD-L1 was found to be involved in tumour-associated immune suppression and host immune damage, thereby promoting cancer progression and subsequent adverse clinical out- comes[3]. In addition, high level of sPD-L1 maybe also associated with the prognosis of malignancies, including colorectal cancer PD-L1, an immune-regulatory molecule, is highly expressed on tumor cells and can be present on activated T and B cell dendritic cells (4). The activation of the programmed death protein 1/programmed death ligand 1 (PD-1/PD-L1) pathway was found as one of the key mechanisms in tumor immune evasion (5). Thus, antibody- based immunotherapies blockading the PD-1/PD-L1 signaling pathways in the tumor microenvironment and stimulating the T-cell anti-tumor activity are a promising approach for developing novel tumor therapeutics in routine clinical practices.

ELIGIBILITY:
Inclusion Criteria:Patients at South Egypt Cancer institute and Assuit University Hospital Recently diagnosed as colorectal cancer patients at different stages.

2. Patients did not undergo colorectal surgery

-

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Cases and controls will be recruited from clinical pathology department at South Egypt Cancer Institute, and Assuit University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Study the expression level of sPDL 1 in colorectal cancer by ELISA | baseline
  Correlate the expression level of sPDL-1 and stage of disease

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shao W, Xu Y, Lin S, Gao J, Gao J, Wang H. The potential of soluble programmed death-ligand 1 (sPD-L1) as a diagnosis marker for colorectal cancer. Front Oncol. 2022 Aug 16;12:988567. doi: 10.3389/fonc.2022.988567. eCollection 2022. PMID 36052227